CLINICAL TRIAL: NCT06211127
Title: Assessment the Safety and Efficacy of Cold Laser Plaque Ablation for Lower Limb Arterial Stenosis and Occlusive Lesions: A Prospective, Multicenter, Randomized Controlled Study.
Brief Title: Safety and Efficacy of Cold Laser Plaque Ablation for Lower Limb Arterial Stenosis and Occlusive Lesions
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Collaborators: First Affiliated Hospital Xi'an Jiaotong University (Other); Henan Provincial People's Hospital (Other); Shanghai Ninth People's Hospital Affiliated to Shanghai Jiao Tong University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZKRG-PAD-202304
Record Dates: First submitted 2023-12-19; First posted 2024-01-18 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2023-12

CONDITIONS: Arterial Disease of Legs; Atherosclerosis of Artery
Keywords: cold laser plaque ablation; lower limb arterial stenosis; occlusive lesions; Atherectomy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cold laser plaque ablation group (Experimental): The disposable cold laser plaque ablation catheter (hereinafter referred to as the ablation catheter) is used in conjunction with the cold laser plaque ablation System), which is suitable for the treatment of arteriosclerosis stenosis and occlusive lesions of the lower limbs.
  Interventions: Device: Cold laser plaque ablation
- The excimer laser group (Active Comparator): Excimer laser uses 308nm wavelength excimer laser to conduct atherosclerotic plaques through the intertwined optical fibers in the catheter, using three action mechanisms of photothermal energy, photochemical energy and acoustic mechanical energy.
  Interventions: Device: The excimer laser

INTERVENTIONS:
Device: Cold laser plaque ablation — Patients were randomly divided into two groups. After being included in the two groups, different laser equipment was used to revascularize the lower limbs. The patients' revascularization status was evaluated through regular follow-up after surgery.
  Arms: Cold laser plaque ablation group
Device: The excimer laser — Patients were randomly divided into two groups. After being included in the two groups, different laser equipment was used to revascularize the lower limbs. The patients' revascularization status was evaluated through regular follow-up after surgery.
  Arms: The excimer laser group

SUMMARY:
This study is a prospective, multi-center, randomized controlled study, which evaluates the effectiveness and safety of cold laser plaque ablation for lower limb arterial stenosis and occlusive lesions from intermittent claudication to chronic threatening limb ischemia.

DETAILED DESCRIPTION:
This study is a prospective, multi-center, randomized controlled study. This study will be conducted at four centers and is expected to enroll 110 patients. And we will evaluate the effectiveness and safety of cold laser plaque ablation compared to excimer laser system for lower limb arterial stenosis and occlusive lesions.

ELIGIBILITY:
Inclusion Criteria:

General selection criteria

1. Age between 18 and 85, gender is not limited;
2. Patients with symptomatic lower extremity arteriosclerosis disease (LEAD), Rutherford grade 2 to 5;
3. The stenosis of lower extremity arteries is greater than 70% or occlusion;
4. The subject is able and willing to comply with all requirements, including 6-month follow-up and evaluation, voluntary participation and informed consent.

Intraoperative contrast inclusion criteria

1. The internal diameter of the reference vessel proximal to the target lesion is greater than 1.8mm;
2. The stenosis of target lesion is greater than 70%;

Exclusion Criteria:

1. The target lesion is located in the artificial vascular or autologous venous vascular bypass;
2. Endovascular or surgical procedure in the target limb performed less than or equal to 30 days prior to the index procedure OR Planned endovascular or surgical procedure 30 days after the index procedure;
3. Intent to use other atherectomy device in the same procedure;
4. Flow-limiting dissection within, proximal or distal to the target lesion;
5. Evidence or history of aneurysm in the target vessel， intracranial or gastrointestinal bleeding, intracranial aneurysm, myocardial infarction or stroke within the past 2 months;
6. Uncorrected coagulation abnormalities (platelet count ≤ 75*109/ L or INR≥2.0), bleeding constitution, and history of heparin-induced thrombocytopenia (HIT);
7. Any thrombolytic therapy was performed within 2 weeks before surgery;
8. History of severe trauma, fracture, major surgery, or parenchymal organ biopsy within 2 weeks before surgery;
9. Known allergy to contrast agents or perioperative drugs;
10. Anticoagulation, antiplatelet or thrombolytic therapy is prohibited;
11. Pregnant or lactating women;
12. Subjects participating in other clinical trials of drugs or medical devices;
13. Other circumstances assessed by the investigator as inappropriate to participate in the trial.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2023-10-16 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
residual diameter stenosis | 1 month, 6 months after surgery
  Reduction from baseline in residual diameter stenosis (measured in percent), prior to any adjunctive therapy, achieved by the laser catheter, as assessed quantitatively by the core laboratory based upon the procedure angiograms.

SECONDARY OUTCOMES:
Secondary effectiveness evaluating indicator:1）Primary patency rate | 1 month, 6 months after surgery
  Proportion of patients with residual vessel diameter greater than 30% within 1 month and 6 months
Secondary effectiveness evaluating indicator:2）Revascularization rate of target vessels | 1 month, 6 months after surgery
  Proportion of patients requiring reoperation for revascularization within 1 month and 6 months due to recurrence or worsening of symptoms caused by the original diseased vessel
Secondary effectiveness evaluating indicator:3）Rutherford grade | 1 month, 6 months after surgery
  Rutherford classification can effectively evaluate the blood supply of patients' lower limbs
Secondary effectiveness evaluating indicator:4）Ankle-brachial index | 1 month, 6 months after surgery
  Ankle-brachial index is generally the ratio of ankle systolic blood pressure to brachial artery systolic blood pressure. Ankle-brachial index is a test method to objectively determine the severity of limb ischemia
Secondary effectiveness evaluating indicator:5)Instrument performance evaluation | 1 month
  Differences in the ablation effects of cold laser and excimer laser on lesions of different nature (thrombus, calcified plaque)
safety evaluating indicator:1) Major Adverse Event (MAE) | 1 month, 6 months after surgery
  Including limb amputation and death due to inversion of diseased blood vessels
safety evaluating indicator:2）Device-associated composite endpoint (Do CE) | 1 month
  Intraoperative device-induced distal embolization or postoperative vascular occlusion
safety evaluating indicator:3）Adverse events / Serious adverse events (AE / SAE) | 1 month, 6 months after surgery
  Adverse events of perforation, dissection, and postoperative hematoma
safety evaluating indicator:4）Incidence of device defects | 1 month
  For example, lesions in certain specific parts cannot be completely removed, etc.

CONTACTS AND LOCATIONS:
Overall Officials: Lianrui Guo, M.D., Study Chair — Xuanwu Hospital, Beijing
Locations (1):
- Xuanwu Hospital, Capital Medical University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No